CLINICAL TRIAL: NCT05696795
Title: JAK1 Inhibition in Sarcoidosis: an Opportunity for Pathogenesis Directed Therapy
Brief Title: Janus Kinase Inhibition in Sarcoidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, William Damsky, Assistant Professor in Dermatology and Dermatopathology, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000033314; 000 (Other: CTGTY)
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Sarcoidosis
Keywords: abrocitinib; JAK1 inhibitor; sarcoidosis
MeSH Terms: conditions — Sarcoidosis | interventions — abrocitinib

STUDY DESIGN:
Intervention Model Description: Male and female subjects at least 18 years of age with moderate to severe cutaneous sarcoidosis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abrocitinib 200 mg daily (Experimental): 6 months of treatment with abrocitinib 200 mg daily
  Interventions: Drug: Abrocitinib 200 mg

INTERVENTIONS:
Drug: Abrocitinib 200 mg — Abrocitinib (Cibinqo) is FDA approved at 200 mg dose once daily for the treatment of atopic dermatitis. It is not currently FDA approved for the treatment of sarcoidosis.

SUMMARY:
The purpose of this study is to investigate the role of the oral JAK1 inhibitor, abrocitinib 200 mg once daily, for the treatment of patients with moderate to severe cutaneous sarcoidosis.

DETAILED DESCRIPTION:
To determine if JAK1 specific inhibition is effective in treating sarcoidosis, an inflammatory condition that can cause disfiguring skin lesions. The only FDA approved therapy is prednisone, a nonspecific immunosuppressant. The primary outcome will be the percent change in the Cutaneous Sarcoidosis Activity and Morphology Instrument (CSAMI) after 6 months of abrocitinib 200 mg daily in 10 patients with moderate to severe cutaneous sarcoidosis.The primary objective of this study is to determine whether oral abrocitinib reduces the CSAMI (a cutaneous sarcoid clinical scoring tool) in patients with moderate to severe cutaneous sarcoidosis. The CSAMI tool was selected over other scoring metrics given the highest interrater reliability of this metric in cutaneous sarcoidosis and the ability to generate subscores for active disease versus scarring. Secondary outcomes will include percent changes in organ involvement on whole body PET-CT imaging, Patients reported outcomes 1) Sarcoidosis related quality-of-life (QoL) metric (King's Sarcoidosis Questionnaire), 2) Skin related quality of life (Skindex-16) metric, 3) sarcoidosis Fatigue Assessment Scale (FAS), and 4) Rhinosinusitis Disability Index (RSDI). Secondary outcomes will also include evaluation of molecular signatures before and during treatment. Soluble IL-2 receptor levels in plasma are the most reliable known biomarker for sarcoidosis and will be assessed at 0 and 6 months. Additional secondary outcomes will include correlative immunologic changes in skin tissue and blood as a result of treatment. Documentation of any spontaneously reported adverse events will be completed throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent.
2. Male and female patients age 18 years old or older.
3. Diagnosis of moderate to severe cutaneous sarcoidosis (CSAMI of 10 or greater) with supportive skin biopsy in which other causes of granulomas (infectious, foreign body) have been ruled out.
4. Patients with either:

   1. Cutaneous Sarcoidosis Activity and Morphology (CSAMI) activity score greater than or equal to 10 (patients with a CSAMI greater than or equal to 10 have active cutaneous sarcoidosis involving several distinct cutaneous sites, have moderate to severe disease and would otherwise be considered candidates for systemic therapy), or
   2. any CSAMI score and skin involvement causing functional impairment (i.e. nasal or visual field obstruction)
5. If patients are taking other systemic therapies for their sarcoidosis, they must be taking a stable dose of the other medication(s) for at least 3 months with no plans to change the regimen in the next 6 months. With the exception of methotrexate or low dose prednisone (20 mg or less per day), use of concomitant immunosuppressants, e.g. infliximab, azathioprine, etc., will not be permitted.

   1. Washout of topical medications will be for 2 weeks.
   2. Washout for oral medications will not be possible in most cases. Patients will be allowed to continue concomitant prednisone (up to 20 mg daily) or weekly methotrexate (up to 15 mg daily).
6. Females of childbearing potential must agree to use birth control during the study and there must be a negative pregnancy test documented prior to starting the medication.
7. Patients must be willing to have skin biopsies, blood collection, and total body photography and to comply with clinic visits.

Exclusion Criteria:

1. Age <18 years old.
2. Patients with a history of malignancy (except history of successfully treated basal cell or squamous cell carcinoma of the skin).

   a) Cutaneous Sarcoidosis Activity and Morphology (CSAMI) activity score less than or equal to 10 or
3. Patients known to be HIV or hepatitis B or C positive, or have an active, serious infection herpes simplex, herpes zoster, and pneumonia. This would also include localized infections as per what is reflected in their medical records.
4. Patients diagnosed with Rheumatoid Arthritis (RA).
5. Patients with positive tuberculin skin test or positive QuantiFERON TB test.
6. Patients with significant hepatic impairment (i.e., Child Pugh C).
7. Patients with moderate to severe renal impairment.
8. Patients with uncontrolled peptic ulcer disease.
9. Patients with advanced or untreated malignancy with the exception of treated non-melanoma skin cancer.
10. Patients with a history of deep vein thrombosis and/or pulmonary embolism and/or clotting disorder.
11. Patients taking immunosuppressive medications, with the exception of methotrexate (up to 20 mg weekly allowed) and/or low-dose prednisone (up to 20 mg daily allowed), including but not limited to mycophenolate mofetil, azathioprine, tacrolimus, cyclosporine, or TNF-α inhibitors.
12. Women of childbearing potential who are unable or unwilling to use birth control while taking the medication.
13. Women who are pregnant or nursing.
14. Current smoker or history of any tobacco use.
15. Screening labs outside the normal range for parameters associated with potential risk for treatment under investigation. Including but not limited to:

    1. Platelets <150,000/mm3
    2. Absolute neutrophil count <1,000/mm3
    3. Hemoglobin levels <8 g/dL
    4. Absolute Lymphocyte Count <300/mm3
16. Patients with any medical, psychiatric or social condition that is likely to unfavorably affect the risk-benefit of continued study participation, interfere with study compliance or confound safety or efficacy assessments.
17. Patients who are taking moderate to strong inhibitors of both CYP2C19 and CYP2C9, or strong CYP2C19 or CYP2C9 inducers, as well as P-gp substrate where small concentration changes may lead to serious or life-threatening toxicities.
18. Patients who have recently received a live vaccine. Patients should wait a minimum of 2 weeks, if recently vaccinated, prior to initiating treatment and should not receive a live vaccine during treatment or 2 weeks post-treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-23 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Changes in Cutaneous Sarcoidosis Activity and Morphology Instrument (CASMI) score | Baseline and 6 Months
  Improvement in the Cutaneous Sarcoidosis Activity and Morphology Instrument (CSAMI) after 6 months of abrocitinib therapy. CSAMI is a validated clinical scoring tool for cutaneous sarcoidosis activity and severity. Scores range from 0 to 165. Higher score is worse.

SECONDARY OUTCOMES:
Percent Changes in Improvement in Internal Organ Involvement | Baseline and 6 Months
  Internal organ involvement and activity will be determined using whole-body positron emission tomography - computed tomography (PET-CT) at baseline and after 6 months of treatment. Change in active inflammation in internal organs will be assessed by calculating total lesion glycolysis (TLG) in affected internal organs. Scores range from 0 to [no upper limit]. Higher score is worse.
Changes in Patient Reported Outcomes Quality of Life (King's Sarcoidosis Questionnaire) | Baseline and 6 Months
  This tool assesses overall quality of life related to sarcoidosis through a questionnaire. Scores range from 1 to 100. Higher score is better.
Changes in Skin related quality of life (Skindex-16) | Baseline and 6 Months
  Skindex-16 is a validated quality of life metric which assesses the effect of diseases involving the skin on individuals' quality of life. It is assessed using a questionnaire. Scores range from 0-96. Higher score is worse.
Changes in Fatigue Assessment Scale (FAS) | Baseline and 6 Months
  FAS is a validated quality of life metric which assesses the effect of sarcoidosis on fatigue / energy level. It is assessed using a questionnaire. Scores range from 0 to 50. Higher score is worse.
Changes in Rhinosinustitis Disability Index (RSDI) | Baseline and 6 months
  RSDI is a validated quality of life metric which assesses the effect sarcoidosis-related nasal sinus symptoms on quality of life. It is assessed using a questionnaire. Scores range from 0 to 120. Higher Score is worse.

CONTACTS AND LOCATIONS:
Overall Officials: William Damsky, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No